CLINICAL TRIAL: NCT04019405
Title: Assessment of Frailty in Elderly People With Ischemic Heart Disease Being Considered for Revascularisation.
Brief Title: Assessing Frailty in Elderly Patients Who Have Ischemic Heart Disease
Acronym: FRAIL_HEART
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 193997
Record Dates: First submitted 2016-10-11; First posted 2019-07-15 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Frail Elderly
Keywords: coronary artery disease; elderly; revascularisation; frailty
MeSH Terms: conditions — Coronary Artery Disease; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Frailty status: Frailty status will be determined by prespecified assessment tools in the study protocol. These assessment tools will be Fried Frailty phenotype model and edmonton frailty Scale.

SUMMARY:
Participants aged 80 years or over, who attend Castle Hill Hospital with either stable angina or an acute coronary syndrome will be invited to participate in the study. After induction into the study, these participants will be assessed for frailty and quality of life (QoL) using predetermined assessment tools. Quality of life (QoL) will be assessed using the standardised SF-12 questionnaire proforma. Frailty assessment will be based on the use of the Fried Frailty Phenotype criteria and the Edmonton Frailty Scale. Patients will be reassessed at 3,9 and 24 months for their clinical outcomes, repeat frailty assessment and quality of life.

DETAILED DESCRIPTION:
STUDY SETTINGS: Cardiology and cardiothoracic out-patients and in-patient wards of Castle Hill hospital

SAMPLE SIZE CALCULATION: FRAIL-HEART is a preliminary observational study designed to evaluate the practicality of undertaking frailty assessments in this population. The sample size of n=150 is estimated on the basis of feasibility. Investigators aim to recruit all consecutive patients who attend our department over a 1 year period. With an expected drop-out rate of 10% , investigators anticipate that it will be feasible to enrol 150 patients in the required time-frame.

PARTICIPANTS: The study target population will be patients aged 80 years or more, who are admitted or referred to the cardiology department because of underlying coronary artery disease.

IDENTIFICATION & RECRUITMENT: These participants will be recruited into the study from outpatient cardiology clinics and from identification of suitable inpatients admitted to the cardiology and cardiothoracic units.

BASELINE ASSESSMENT: The baseline assessment will include gathering patient baseline demographic data, current diagnosis and clinical status, assessment of the comorbid conditions, and information regarding relevant investigation results including blood results, electrocardiogram (ECG), echocardiogram and coronary angiography data. Participants will be asked to complete QoL questionnaire and undergo the frailty assessments. This will entail completion of several questionnaires.

SF-12 QoL QUESTIONNAIRE: This questionnaire of 12 questions have been extensively used in research practice and validated to assess QoL in a variety of clinical settings20.

FRAILTY ASSESSMENT: This will be evaluated using both the Fried phenotype and Edmonton frailty scale. Study participants will first be asked to complete the written questionnaires. They will then have a measure of handgrip strength and if feasible will be asked to do 'get up and go' and 'five metre walk 'test as detailed in the Edmonton and Fried assessments respectively. Participants who are unable to walk will be marked as per the criteria. Where applicable, participants will be allowed to use walking aids as required.

Where applicable, the research team will also evaluate the results of coronary angiography and will undertake both SYNTAX as well as EUROSCORE calculations.

FOLLOW UP ASSESSMENTS: The study participants will be seen at 3, 9 and 24 month intervals and will be asked to complete the QoL questionnaire and undergo frailty assessment. The following variables will be recorded at each follow-up visit.

* Patient symptoms- CCS angina class, NYHA class
* Height, weight, BMI, Vital signs
* Medication with dosages
* Document all major adverse outcomes: myocardial infarction, acute cerebrovascular event, major bleeding, or unplanned re-hospitalisation.
* Document any other adverse events such as kidney injury, transient ischaemic attack.
* Document length of stay on ICU and total length of hospital stay (where applicable).
* SF-12 questionnaire
* Fried Frailty phenotype
* Edmonton frailty scale
* Patient perspective survey form- Two separate patients perspective have been developed depending whether the study participants are managed medically or undergo intervention and cardiac surgery.

DEATHS DURING THE STUDY PERIOD: Due to the advanced age of the study participants, it is expected that some patients might die during the study period. In such a situation the data already gathered will be retained in the study. Investigators will be advised to check on the Hull and East Yorkshire NHS Trust record systems before sending out any follow up appointments. The participant's family and relatives will not be approached after their death.

ELIGIBILITY:
Inclusion Criteria:

Aged 80 years and above and either

1. Have been seen in the cardiology out-patient department with a diagnosis of stable angina
2. Have been admitted to Castle Hill Hospital with non-ST elevation acute myocardial infarction (NSTEMI)
3. Have been admitted to Castle Hill Hospital with ST-elevation acute myocardial infarction (STEMI)
4. Have been referred to Castle Hill Hospital for coronary angioplasty
5. Have been referred to Castle Hill Hospital for coronary artery bypass graft surgery

Exclusion Criteria:

Patients will be excluded from the study in the event of any of the following:

1. Patients who are unable to provide informed consent including those with advanced dementia.
2. Patients, who are not able to speak good English sufficiently to be able to understand the study information, give consent and complete study measures.
3. Patients who have a primary diagnosis of significant valvular disease

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients (male and female) aged 80 and over and who have a primary diagnosis of ischaemic heart disease will be eligible for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Quality Of Life Questionnaire | baseline and 3, 9 and 24 months
  The primary out come will be quality of life assessed by SF-12 survey forms

SECONDARY OUTCOMES:
Change in frailty Status - Fried frailty Criteria | baseline and 3, 9 and 24 months
  To evaluate changes in frailty using the Fried frailty criteria.
Change in frailty Status - Edmonton Frailty Score | baseline and 3, 9 and 24 months
  To evaluate changes in frailty using the Edmonton frailty score.
Major adverse clinical events during hospitalization | baseline and 3, 9 and 24 months
  To evaluate major adverse clinical event (MACE) (defined as a composite of death, acute myocardial infarction, acute cerebrovascular event (CVA), and major bleeding) occurring during hospitalisation for frail versus non-frail participants of study.
Major Adverse Clinical Event | 24 months
  To evaluate major adverse clinical event (MACE) (defined as a composite of death, acute myocardial infarction, acute cerebrovascular event (CVA), major bleeding, and unplanned rehospitalisation occurring at 24 months follow-up for frail versus non-frail participants of the study.
Predictors of adverse outcome | baseline and 3, 9 and 24 months
  Patients' variables will be evaluated to determine the independent predictors of an adverse outcome (defined as death or a worsening in QOL at follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hoye, MB.ChB,PhD, Principal Investigator — Hull and East Yorkshire NHS Trust
Locations (1):
- Castle Hill Hospital, Cottingham, East Riding of Yorkshire NHS Trust, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared